CLINICAL TRIAL: NCT00736255
Title: Lis-dexamphetamine (LDX/SPD489)as a Treatment for Smoking Cessation in Nicotine Dependent Individuals With ADHD
Brief Title: Attention Deficit Hyperactivity Disorder (ADHD) Smoking Cessation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Shire (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00001248; SPD489-607 (Other Grant/Funding Number: Shire Pharmaceuticals)
Record Dates: First submitted 2008-08-13; First posted 2008-08-15 (Estimated); Results first posted 2012-09-07 (Estimated); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Attention Deficit Hyperactivity Disorder; Nicotine Dependence
Keywords: ADHD; Smoking
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Tobacco Use Disorder; Smoking | interventions — Tobacco Use Cessation Devices; Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vyvanse and transdermal nicotine patch (Experimental): The first group will receive LDX/SPD489 titrated up to 70 mg qd for 4 weeks after the identified quit date. Subjects will continue to receive NRT 21 mg at week 1 post quit date, then 14mg at week 2 post quit date and 7 at weeks 3 and 4 post quit date.
  Interventions: Drug: Transdermal Nicotine Patch; Drug: Lis-dexamphetamine (Vyvanse)
- Placebo and transdermal nicotine patch (Placebo Comparator): The second group will receive matching placebo and NRT after the quit date.
  Interventions: Drug: Transdermal Nicotine Patch; Drug: Placebo

INTERVENTIONS:
Drug: Transdermal Nicotine Patch — All subjects will lreceive transdermal nicotine patch during beginning at Visit 0 (quit smoke date). The dose will be tapered down from 21 mg to 14mg after week 1,vthen to 7 mg after week 2. Subjects will remain at 7mg until the 4th week.
  Other Names: Nicotine Patch
Drug: Lis-dexamphetamine (Vyvanse) — Subjects on this arm will receive Lis-dexamphetamine day after the identified quit date. All subject will start with 30mg once a day and will be titrated up to 50mg then to 70mg over a 3 week period to reach an optimized dose. They will then be maintained on this optimized dose until the 4th week.
  Other Names: LDX and Transdermal Nicotine Patch
  Arms: Vyvanse and transdermal nicotine patch
Drug: Placebo — Subjects on this arm will receive matching placebo, along with Nicotine Replacement Therapy.
  Other Names: Placebo and Transdermal Nicotine Patch
  Arms: Placebo and transdermal nicotine patch

SUMMARY:
The overall goal of the present project is to investigate whether lisdexamphetamine (LDX; Vyvanse) is an effective adjunct to nicotine replacement therapy (NRT) to promote smoking cessation in patients with comorbid Attention Deficit Hyperactivity Disorder (ADHD) and nicotine dependence. The investigators hypothesized initially that smokers with ADHD who are optimized to a dose of LDX prior to quitting smoking and who remain on this dose of medication after quitting will remain abstinent longer than patients who are treated with placebo before and after quitting.However due to recent key issues that have arisen showing that initiation of stimulant treatment while subjects are actively smoking may facilitate increased smoking, and given that the study was still in the very early stage of study execution, the investigators revised the study design to use an empirically validated pretreatment approach with NRT and to initiate LDX treatment on the first post quit date in order to reduce the withdrawal symptoms that accompany smoking cessation. The overall rationale for this revised study design remains similar to the original.

DETAILED DESCRIPTION:
This will be a 2-group, parallel, placebo-controlled, double blind study. Regular, nicotine dependent individuals with ADHD will receive NRT pretreatment for 2 weeks prior to an identified quit date.At the quit date, subjects will be randomized into one of two groups.

* The first group will begin treatment for 1 week with LDX 30 mg and then will be titrated up to 50mg and 70mg if tolerated. Subjects will continue on the highest tolerated dose until the 4th week. Concurrently subjects will receive transdermal NRT, 21 mg at week one, 14 mg at week 2 and 7 mg at weeks 3 and 4.
* The second group will receive matching placebo and transdermal NRT after the quit date.

Participants will attend a total of 16 visits over a period of 7-11 weeks. The primary outcome measure for this study will be the proportion of individuals in each group who report 4 weeks continuous smoking abstinence verified by both Carbon Monoxide (CO) levels and salivary cotinine, measured at Visit 5. It is hypothesized that the group co-treated with LDX will have a significantly higher proportion of individuals who remain abstinent across the 4 weeks measured every other day.

Inclusion Criteria:

* Aged 18-50 years
* Meet DSM-IV criteria (Diagnostic and Statistical manual of mental Disorders Version 4) for ADHD, any subtype; assessed using the Conners Adult ADHD Interview for DSM (CAADID)
* Meet DSM-IV criteria for nicotine dependence as verified by afternoon expired CO levels of >15 parts per million (PPM) and self-report of smoking >10 cigarettes/day
* Free from major medical problems and deemed healthy by the study physician
* Not currently receiving medication for ADHD or other psychiatric disorders. If a patient is screened as is currently receiving medication for ADHD, they may be enrolled, provided they washout of their current medication for an appropriate length of time.
* No contraindications for treatment with either LDX or transdermal nicotine

Exclusion Criteria:

* DSM-IV Axis I or Axis II disorders that require additional pharmacological treatment or otherwise would interfere with participation in the present study
* History of known cardiovascular disease, clinically significant hypertension, or other cardiovascular risk factors which, in the opinion of the study physician, would contraindicate treatment
* BMI (Body Mass Index) > 35

ELIGIBILITY:
Inclusion Criteria:

* Attention Deficit Hyperactivity Disorder(ADHD) diagnosis
* smokes at least > 10 cigarettes per day
* no major medical problems
* no contraindications to treatment with either LDX or transdermal nicotine

Exclusion Criteria:

* other psychiatric conditions that require medication
* history of cardiovascular disease, clinically significant hypertension
* Body Mass index (BMI) > 35

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2007-12; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott H Kollins, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Attention Deficit Hyperactivity Disorder (ADHD) Program, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment ended in March 2011 at the Duke.A total of 59 subjects were screened. 24 did not pass screening while 35 were eligible. Of the 35 screen passers, 32 were randomized to receive either LDX or placebo, 3 were withdrawn prior to randomization. Of the 32 randomized, 17 received LDX and 15 received placebo. 14 completed on each arm.
Pre-assignment Details: There were 24 screen fails. Reason for Screen Fails include:Did not complete screening - 2,Carbon monoxide too low - 3,Positive Urine drug screen - 3,Physical health reasons - 5,Psychiatric comorbidity - 11
Groups:
- LDX and NRT: • The first group will receive LDX/SPD489 titrated up to 70 mg qd for 4 weeks after the identified quit date. Subjects will continue to receive NRT 21 mg at week 1 post quit date, then 14mg at week 2 post quit date and 7 at weeks 3 and 4 post quit date.
- NRT and Placebo: The second group will receive matching placebo and NRT after the quit date.
Period: Overall Study
Arm/Group | LDX and NRT | NRT and Placebo
Started | 17 | 15
Completed | 14 | 14
Not Completed | 3 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Non-compliance | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LDX and NRT | NRT and Placebo | Total
Number analyzed (Participants) | 17 | 15 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 15 | 32
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.6 (8.4) | 33.5 (9.1) | 31 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 11 | 6 | 17
Region of Enrollment [Number; unit: participants]
  United States | 17 | 15 | 32

OUTCOME MEASURES:

1. Primary Outcome: The Number of Subjects in Each Treatment Group Exhibiting Sustained, 4-week Smoking Abstinence, Defined as CO Levels <= 4 Ppm for Each Post-quit Study Visit.
Description: The primary outcome measure was the proportion of subjects in each treatment group exhibiting sustained, 4-week smoking abstinence, defined as CO levels <= 4 ppm for each post-quit study visit. Subjects who dropped from the study for any reason were considered to have lapsed.
Time Frame: 4 weeks
Population: Subjects exhibiting sustained 4 week smoking abstinence defined as CO levels <= 4ppm for each post quit study visit were analyzed for the outcome measure.
Measure: Number; unit: participants
Groups:
- LDX and NRT: • The first group will receive LDX/SPD489 titrated up to 70 mg qd for 4 weeks after the identified quit date. Subjects will continue to receive NRT 21 mg at week 1 post quit date, then 14mg at week 2 post quit date and 7 at weeks 3 and 4 post quit date.
  Lis-dexamphetamine (LDX; Vyvanse) and Transdermal Nicotine Patch: Subjects on this arm will receive Lis-dexamphetamine day after the identified quit date. All subject will start with 30mg once a day and will be titrated up to 50mg then to 70mg over a 3 week period to reach an optimized dose. They will then be maintained on this optimized dose until the 4th week. All subjects will continue to receive transdermal nicotine patch during these weeks. The dose will be tapered down from 21 mg to 14mg after week 1,then to 7 mg after week 2. Subjects will remain at 7mg until the 4th week.
- NRT and Placebo: The second group will receive matching placebo and NRT after the quit date.
  Placebo and transdermal nicotine patch: Subjects on this arm will receive matching placebo and NRT.
Arm/Group | LDX and NRT | NRT and Placebo
Number analyzed (Participants) | 17 | 15
participants | 5 | 3
Statistical Analysis 1: Comparison: LDX and NRT vs NRT and Placebo; Null Hypothesis:LDX and NRT will not facilitate smoking cessation compared to NRT and placebo. Alternate Hypothesis: LDX and NRT will facilitate smoking cessation compared to NRT and placebo. This is a one tailed, proof of concept study so there is no formal power analysis, however if we see a signal for treatment effect, we would like to do further investigation by conducting a separate trial; Test type: Superiority or Other; p = 0.54, Chi-squared

2. Secondary Outcome: Smoking Rates
Description: Smoking rates, measured as self-reported cigarettes/day.
Time Frame: Randomization, visits 1 (day 4), 2 (day 7), 3 (day 11), 4 (day 14), 5 (day 18), 6 (day 21), 7 (day 25), 8 (day 28)
Measure: Mean (Standard Error); unit: Cigarettes smoked per day
Arm/Group | LDX and NRT | NRT and Placebo
Number analyzed (Participants) | 17 | 15
Cigarettes smoked per day
  Randomization (Visit 0) | 6.43 (1.38) | 8.14 (1.79)
  Visit 1 (day 4) | 3.90 (1.28) | 2.59 (1.02)
  Visit 2 (day 7) | 3.16 (1.10) | 1.83 (0.84)
  Visit 3 (day 11) | 2.75 (1.12) | 2.23 (0.94)
  Visit 4 (day 14) | 2.98 (1.31) | 2.10 (0.74)
  Visit 5 (day 18) | 3.08 (1.45) | 2.92 (1.00)
  Visit 6 (day 21) | 3.94 (1.59) | 2.67 (0.98)
  Visit 7 (day 25) | 4.38 (1.69) | 2.33 (0.84)
  Visit 8 (day 28) | 4.15 (1.58) | 2.91 (1.07)

3. Secondary Outcome: Continuous Performance Test (CPT) Commission Errors
Description: The CPT is a measure of both vigilance/sustained attention and response inhibition, has good normative data and has been shown to be sensitive to the effects of stimulants. Reaction time variability and commission errors - measures of attentional control and response inhibition have been shown to be sensitive in discriminating individuals with ADHD on active medication versus placebo.
Time Frame: Randomization, Visits 1 (day 4), 2 (day 7), 3 (day 11), 4 (day 14), 5 (day 18), 6 (day 21), 7 (day 25), 8 (day 28)
Measure: Mean (Standard Deviation); unit: Errors of Commission
Arm/Group | LDX and NRT | NRT and Placebo
Number analyzed (Participants) | 17 | 15
Errors of Commission
  Randomization (Visit 0) | 15.29 (10.58) | 12.43 (9.37)
  Visit 1 (day 4) | 13.29 (9.64) | 10.71 (8.62)
  Visit 2 (day 7) | 13.44 (9.14) | 10.86 (8.70)
  Visit 3 (day 11) | 14.50 (8.91) | 10.79 (7.52)
  Visit 4 (day 14) | 13.13 (8.33) | 11.08 (9.29)
  Visit 5 (day 18) | 15.00 (7.67) | 11.15 (9.20)
  Visit 6 (day 21) | 12.36 (10.43) | 12.15 (8.12)
  Visit 7 (day 25) | 14.64 (9.20) | 11.77 (6.98)
  Visit 8 (day 28) | 14.92 (10.80) | 11.23 (9.77)

4. Secondary Outcome: Continuous Performance Test (CPT) Reaction Time Standard Error
Description: as for outcome 3
Time Frame: Randomization, Visits 1 (day 4), 2 (day 7), 3 (day 11), 4 (day 14), 5 (day 18), 6 (day 21), 7 (day 25), 8 (day 28)
Measure: Mean (Standard Deviation); unit: Reaction time in seconds
Arm/Group | LDX and NRT | NRT and Placebo
Number analyzed (Participants) | 17 | 15
Reaction time in seconds
  Randomization (Visit 0) | 5.37 (1.93) | 4.61 (1.31)
  Visit 1 (day 4) | 5.52 (3.44) | 4.68 (1.44)
  Visit 2 (day 7) | 5.42 (3.45) | 5.05 (1.81)
  Visit 3 (day 11) | 4.97 (2.71) | 5.01 (1.46)
  Visit 4 (day 14) | 4.83 (2.55) | 4.79 (1.71)
  Visit 5 (day 18) | 5.54 (2.77) | 5.15 (1.71)
  Visit 6 (day 21) | 4.64 (2.28) | 4.97 (1.62)
  Visit 7 (day 25) | 5.29 (2.73) | 5.73 (2.01)
  Visit 8 (day 28) | 4.86 (2.23) | 5.08 (2.04)

5. Secondary Outcome: ADHD Conners' Adult ADHD Rating Scales (CAARS) Self-Report and Observer Short Forms
Description: T-scores derived from compiled ADHD symptoms from two forms. Specifically the t-scores for the DSM-IV Total subscale, representing ADHD symptoms. This is conducted by the participant and clinician at randomization, visits 2 and 4 (i.e. dose titration visits), Visit 6 (i.e. monitoring visit), and Visit 8 (i.e. final/end of study visit).
  The following describes severity of the ADHD symptoms (based upon T-Score):
  70+ = Very Much Above Average 66-70 = Much Above Average 61-65 = Above Average 56-60 = Slightly Above Average 45-55 = Average 30-44 = Below Average (Low scores are good)
Time Frame: Randomization, Visits 2 (day 7), 4 (day 14), 6 (day 21), 8 (day 28)
Measure: Mean (Standard Deviation); unit: T-score on a scale
Arm/Group | LDX and NRT | NRT and Placebo
Number analyzed (Participants) | 17 | 15
T-score on a scale
  Randomization (Visit 0) | 67.13 (9.75) | 68.08 (7.48)
  Visit 2 (day 7) | 63.07 (11.48) | 64.62 (8.69)
  Visit 4 (day 14) | 58.62 (13.18) | 65.25 (9.85)
  Visit 6 (day 21) | 52.83 (17.07) | 63.42 (12.70)
  Visit 8 (day 28) | 54.00 (15.33) | 61.92 (11.46)

6. Secondary Outcome: N-back Test Proportion Correct Across 4 Load Factors
Description: This is measured by the N-Back test, a cognitive functioning, including working memory test. The test is designed with 4 Load Factors, where the current stimulus matches the one from 'n' steps back or prior in the sequence. The load factor n is adjusted so there is a 'O-back' (i.e. 'n-0'), '1-back' (i.e. 'n-1'), '2-back' (i.e. 'n-2'), and '3-back' (i.e. 'n-3'). When the correct stimulus appears on the screen, the participant then responds on the computer. Missing the stimulus decreases the proportion correct.
Time Frame: Randomization, Visits 1 (day 4), 2 (day 7), 3 (day 11), 4 (day 14), 5 (day 18), 6 (day 21), 7 (day 25), 8 (day 28)
Measure: Mean (Standard Deviation); unit: proportion correct to stimuli response
Arm/Group | LDX and NRT | NRT and Placebo
Number analyzed (Participants) | 17 | 15
proportion correct to stimuli response
  Randomization (Visit 0) 0-back _%cor | 0.96 (0.12) | 1.00 (0.00)
  Randomization (Visit 0) 1-back _%cor | 0.94 (0.15) | 0.99 (0.03)
  Randomization (Visit 0) 2-back _%cor | 0.96 (0.08) | 0.95 (0.09)
  Randomization (Visit 0) 3-back _%cor | 0.84 (0.14) | 0.80 (0.29)
  Visit 1 (day 4) 0-back _%cor | 0.95 (0.23) | 1.00 (0.00)
  Visit 1 (day 4) 1-back _%cor | 0.90 (0.25) | 0.99 (0.02)
  Visit 1 (day 4) 2-back _%cor | 0.89 (0.27) | 0.96 (0.09)
  Visit 1 (day 4) 3-back _%cor | 0.80 (0.31) | 0.83 (0.18)
  Visit 2 (day 7) 0-back _%cor | 0.93 (0.26) | 0.92 (0.27)
  Visit 2 (day 7) 1-back _%cor | 0.90 (0.26) | 0.95 (0.11)
  Visit 2 (day 7) 2-back _%cor | 0.86 (0.30) | 0.92 (0.13)
  Visit 2 (day 7) 3-back _%cor | 0.81 (0.28) | 0.81 (0.27)
  Visit 3 (day 11) 0-back _%cor | 0.89 (0.27) | 0.99 (0.02)
  Visit 3 (day 11) 1-back _%cor | 0.89 (0.28) | 0.99 (0.02)
  Visit 3 (day 11) 2-back _%cor | 0.89 (0.27) | 0.95 (0.10)
  Visit 3 (day 11) 3-back _%cor | 0.84 (0.30) | 0.90 (0.14)
  Visit 4 (day 14) 0-back _%cor | 0.93 (0.26) | 0.99 (0.02)
  Visit 4 (day 14) 1-back _%cor | 0.91 (0.26) | 0.99 (0.03)
  Visit 4 (day 14) 2-back _%cor | 0.90 (0.25) | 0.95 (0.12)
  Visit 4 (day 14) 3-back _%cor | 0.90 (0.25) | 0.89 (0.15)
  Visit 5 (day 18) 0-back _%cor | 1.00 (0.00) | 0.99 (0.03)
  Visit 5 (day 18) 1-back _%cor | 0.98 (0.08) | 0.99 (0.02)
  Visit 5 (day 18) 2-back _%cor | 0.99 (0.02) | 0.98 (0.08)
  Visit 5 (day 18) 3-back _%cor | 0.88 (0.16) | 0.92 (0.16)
  Visit 6 (day 21) 0-back _%cor | 0.93 (0.27) | 1.00 (0.00)
  Visit 6 (day 21) 1-back _%cor | 0.93 (0.27) | 0.98 (0.03)
  Visit 6 (day 21) 2-back _%cor | 0.90 (0.26) | 0.96 (0.09)
  Visit 6 (day 21) 3-back _%cor | 0.89 (0.26) | 0.87 (0.15)
  Visit 7 (day 25) 0-back _%cor | 0.99 (0.03) | 0.99 (0.04)
  Visit 7 (day 25)1-back _%cor | 0.99 (0.03) | 0.99 (0.03)
  Visit 7 (day 25) 2-back _%cor | 0.97 (0.07) | 0.95 (0.12)
  Visit 7 (day 25) 3-back _%cor | 0.91 (0.11) | 0.88 (0.15)
  Visit 8 (day 28) 0-back _%cor | 0.93 (0.23) | 0.99 (0.02)
  Visit 8 (day 28) 1-back _%cor | 0.98 (0.03) | 0.98 (0.05)
  Visit 8 (day 28) 2-back _%cor | 0.92 (0.27) | 0.95 (0.09)
  Visit 8 (day 28) 3-back _%cor | 0.91 (0.13) | 0.84 (0.21)

7. Secondary Outcome: Clinician Rated Clinical Global Impressions of Improvement Scale (CGI-I)
Description: Measures clinician's perception of patient improvement at the time of assessment compared with the start of treatment. 1-Very Much Improved through 7-Very Much Worse.
Time Frame: Visits 2 (day 7), 4 (day 14), 6 (day 21), 8 (day 28)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LDX and NRT | NRT and Placebo
Number analyzed (Participants) | 17 | 15
score on a scale
  Visit 2 (day 7) CGI-I | 2.88 (0.89) | 3.50 (0.76)
  Visit 4 (day 14) CGI-I | 2.73 (1.03) | 3.38 (0.77)
  Visit 6 (day 21) CGI_I | 2.29 (1.20) | 3.31 (1.18)
  Visit 8 (day 28) CGI-I | 2.00 (1.24) | 3.15 (0.99)

ADVERSE EVENTS:
Arm/Group | LDX and NRT | NRT and Placebo
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/15
Other Adverse Events (participants affected / at risk) | 15/17 | 12/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LDX and NRT (N=17) | NRT and Placebo (N=15)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1)
Inability to concentrate (Psychiatric disorders) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 3 (3) | 1 (1)
Panic Attack (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Nightmares/Dreams (Psychiatric disorders) | 3 (3) | 3 (3)
Increased Appetite (Psychiatric disorders) | 1 (1) | 0 (0)
Decreased Appetite (Psychiatric disorders) | 6 (6) | 1 (1)
Excessive Thirst (General disorders) | 1 (1) | 1 (1)
Chest tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Muscle twitches (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Stomach ache (Gastrointestinal disorders) | 1 (1) | 1 (1)
Arm Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bruxism (Psychiatric disorders) | 2 (2) | 0 (0)
Heartburn (Gastrointestinal disorders) | 0 (0) | 2 (2)
Fatigue (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Shaking hands/Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Nervous system disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 4 (4) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 6 (6)
Chills (General disorders) | 0 (0) | 1 (1)
Skin irritation at NRT patch site (Skin and subcutaneous tissue disorders) | 1 (1) | 7 (7)
Dry mouth (General disorders) | 2 (2) | 0 (0)
Metallic Taste (Endocrine disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations of the study: 1. Our sample size was quite small and this can realistically only be considered a pilot trial. 2.We did not collect systematic follow-up data on our sample after the end of treatment.3.the duration of our trial was short.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No